CLINICAL TRIAL: NCT02791061
Title: Segmentation, Structural Reconstruction and Quantification of Right Ventricular Remodeling in Congenital Heart Disease for Clinical Decision-making and Treatment Planning.
Brief Title: Study of RV Remodeling in Congenital Heart Disease
Acronym: RVShape
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/856/C
Record Dates: First submitted 2016-05-31; First posted 2016-06-06 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: Healthy Volunteers will undergo the following studying procedures:
  Cardiovascular Magnetic Resonance Imagine (MRI) Cardiopulmonary exercise testing (CPET) Echocardiography
  Interventions: Other: Cardiovascular Magnetic Resonance Imagine (MRI); Other: Cardiopulmonary exercise testing (CPET); Other: Echocardiography
- Congenital Disease: Patients will undergo the following studying procedures:
  Cardiovascular Magnetic Resonance Imagine (MRI) Cardiopulmonary exercise testing (CPET) Echocardiography
  Interventions: Other: Cardiovascular Magnetic Resonance Imagine (MRI); Other: Cardiopulmonary exercise testing (CPET); Other: Echocardiography

INTERVENTIONS:
Other: Cardiovascular Magnetic Resonance Imagine (MRI) — MRI uses interaction of the magnetic properties of body tissues with strong magnetic fields to create images.
Other: Cardiopulmonary exercise testing (CPET) — Cardiopulmonary exercise testing (CPET) is non-invasive simultaneous measurement of the cardiovascular and respiratory system during exercise to assess a patient's exercise capacity.
Other: Echocardiography — To measure heart chamber size, heart function, blood vessel size and blood vessel function. These measurements will help us understand the type and severity of heart failure.

SUMMARY:
The primary aims of this study are to 1. Develop an automated method of quantitation of RV remodeling in terms of regional RV surface curvature and area strain and assess the feasibility, repeatability and accuracy in normal subjects and patients with repaired TOF, patients with PS

The secondary study aims of this study are to

1. Compare the differences of RV remodeling in repaired TOF patients, PS patients with sex and age-matched controls 2, Assess the relationship of our proposed parameters to global RV function and exercise capacity in repaired TOF patients and PS patient

DETAILED DESCRIPTION:
Right ventricular (RV) function is increasingly recognized to play an important role in the clinical status and long-term outcome in patients with congenital heart disease (CHD) as well as ischemic cardiomyopathy with left ventricular (LV) dysfunction. However, quantitation of RV characteristics and function, in particular for regional RV characteristics and function, are still challenging due to its complex morphology and its thin wall with coarse trabeculations. The remarkable improvement in survival of CHD patients has led to a continuously growing number of grown-up CHD. In addition, some defects (e.g., Ebstein's anomaly) may be diagnosed for the first time in adult. Majority of these CHD patients face a lifetime of problems including RV dilation, ventricular arrhythmias, and sudden cardiac death. Therefore, accurate depictions of the RV remodeling process facilitate disease would aid in surveillance and monitoring of therapeutic efficacy.

CHD patients, even after corrective surgery, need lifetime surveillance and yearly clinical evaluation. Currently, clinical evaluation includes ECG and pulse oximetries alongside clinical examination. Investigation of anatomy and physiology of RV are changing from invasive studies (right heart catheterization) to noninvasive imaging techniques including: echocardiography, nuclear scintigraphy, computed tomography, and cardiac magnetic resonance (CMR) imaging. In short, echocardiography is largely operator dependent and suffers from poor inter-study reproducibility. The complex geometry of the RV makes it difficult to accurately quantify its remodeling before and after intervention. Nuclear scintigraphy and computed tomography are constrained by the need for ionizing radiation as well as the poor temporal resolution of the technique. CMR has been considered the golden reference technique for RV volume and ejection fraction.

From current state-of-the-art in CMR, generation of RV volume and ejection fraction, global measures of RV remodeling, requires extensive manual contouring. Most important, there is lacking of regional RV remodeling measures.

ELIGIBILITY:
Inclusion Criteria:

1. Survivors of TOF repair more than one year after repair without pulmonary stenosis (Doppler gradient more than 30mmHg) OR
2. Patients with moderate or severe pulmonary stenosis (Echo Doppler gradient more than 30mmHg)
3. Patients without prior Pulmonary Valve Replacement (PVR)
4. Written informed Consent obtained
5. Aged 13 to 80 years old

Exclusion Criteria:

1. Age less than 13
2. Contraindication to MRI Examination

   * Cardiac Pacemaker
   * Brain Aneurysm OR clips
   * Electronic implants OR prosthesis
   * Eye metal foreign body injury
   * Severe claustrophobia
   * Known severe impairment, glomerular filtration rate GFR less than 30 ml/min/BSA
3. Non Cardiac illness with life expectancy of less than 2 years
4. Previous heart kidney liver or lung transplantation Pregnancy

Ages: 13 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 34 patients diagnosed will Tetralogy of Fallots or Pulmonary Stenosis will be recruited from primary care clinic, outpatient clinics and hospital ward in NHCS.
  20 Healthy Volunteer control group.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2013-01; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
First occurrence of cardiovascular event | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Ru San Tan, MBBS, Principal Investigator — National Heart Centre Singapore
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No